CLINICAL TRIAL: NCT02703974
Title: Nudging Handwashing: a Cluster-randomized Trial in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Save the Children (Other); University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 6304
Record Dates: First submitted 2016-02-18; First posted 2016-03-09 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Hand Disinfection
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Early handwashing station + nudge (Experimental): This arm will include 5 randomly selected schools that will have had handwashing stations built after the baseline observation (Phase I), and nudges built after Phase II data collection.
  Interventions: Behavioral: Early handwashing station; Behavioral: Nudge
- Late handwashing station + nudge (Experimental): This arm will include 5 randomly selected schools that will have had handwashing stations and nudges built at the same time, after Phase II data collection.
  Interventions: Behavioral: Late handwashing station; Behavioral: Nudge
- Early handwashing station + education (Active Comparator): This arm will include 5 randomly selected schools that will have had handwashing stations built after the baseline observation (Phase I), and will receive a Hand hygiene education-based program, after Phase II data collection is complete.
  Interventions: Behavioral: Early handwashing station; Behavioral: Education
- Late handwashing station + education (Active Comparator): This arm will include 5 randomly selected schools that will have had handwashing stations built after Phase II data collection is complete, when the Hand hygiene education-based program will commence.
  Interventions: Behavioral: Late handwashing station; Behavioral: Education

INTERVENTIONS:
Behavioral: Early handwashing station — A handwashing station will be a dedicated location for handwashing in each selected school and will include:
  1. A raised concrete platform (built to child height)
  2. A plastic container with a lid and spigot
  3. Soap
  The early handwashing stations will be constructed in weeks 1 and 2 of the study, after the baseline observations (Phase I) are complete.
  Arms: Early handwashing station + education; Early handwashing station + nudge
Behavioral: Late handwashing station — A handwashing station will be a dedicated location for handwashing in each selected school and will include:
  1. A raised concrete platform (built to child height)
  2. A plastic container with a lid and spigot
  3. Soap
  The late handwashing stations construction will begin after Phase 2 data collection has been finished at the end of week 3.
  Arms: Late handwashing station + education; Late handwashing station + nudge
Behavioral: Nudge — A nudge will be built in each randomly selected school and will consist of:
  1. Connecting latrines to the handwashing station via paved pathways that are painted bright colors
  2. Painting footprints on infrastructure guiding students to the handwashing stations and handprints on stations
  The nudges will be constructed at the end of week 3 and 4, after Phase II data collection is complete within each randomly assigned nudge school.
  Arms: Early handwashing station + nudge; Late handwashing station + nudge
Behavioral: Education — Hand hygiene education-based program: the hygiene promotion element will include a one month program of handwashing education involving weekly facilitator led sessions. Each session will be about 30-45 minutes long, and will cover the following topics:
  * Importance of handwashing
  * Method of handwashing
  * Critical times of handwashing
  * Finding solutions for handwashing in school and at home The sessions will involve use of flipcharts, and other IEC materials (e.g. videos) and participative learning methods.
  The Hand hygiene education-based program will begin at the beginning of weeks 4 and 5, after Phase II data collection is complete in each randomly assigned education school.
  Arms: Early handwashing station + education; Late handwashing station + education

SUMMARY:
The study will collect and analyze quantitative data regarding handwashing behaviors among school-aged children to determine the impact of nudges compared to handwashing and hygiene education programs.

Based on the success of the preliminary pilot, we hypothesize nudges leading to higher rates of handwashing than traditional handwashing and hygiene education programs.

DETAILED DESCRIPTION:
This study will utilize a cluster-randomized trial design to collect quantitative data and analyze the handwashing behaviors of school-aged children.

The primary purpose of this protocol is to assess nudges as a viable method of promoting handwashing among school-aged children.

The specific objectives of this quantitative exploration are to:

1. Determine if nudges can prompt significant behavior change and result in higher rates of handwashing among school-aged children in Bangladesh
2. Determine if behavior change resulting from nudging is sustainable over time

ELIGIBILITY:
Inclusion Criteria:

* schools in Dhunat, Gurudaspur and Boraigram Upazilla (sub districts) of Bogra and Natore districts of Rajshahi Division that that meet the following inclusion criteria:

  1. No hygiene education programs in the last two years
  2. No handwashing stations or facilities on school grounds
  3. Improved sanitation/toilets facilities (latrines)
  4. Water supply on site or within 3-6 meters of the school
  5. A school population between 125-450 students, and
  6. A government primary school (all co-ed)
  7. Willingness of the school principle / head teacher and a representative of the School Management Committee (SMC) to participate in the proposed research

Exclusion Criteria:

1. Located outside of Dhunat, Gurudaspur and Boraigram Upazilla (sub districts) of Bogra and Natore districts of Rajshahi Division
2. Have had a hygiene education program in the last two years
3. Already has handwashing stations or facilities on school grounds
4. Does not have improved sanitation/toilets facilities (latrines)
5. Does not have water supply on site or within 3-6 meters of the school
6. Has a school population under 125 or over 450 students
7. Is not a government primary school or is not co-ed
8. School principle / head teacher or representative of the School Management Committee (SMC) is not willing to participate in the proposed research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the probability of handwashing with soap after a toileting event among students receiving nudge intervention compared to that of students in hygiene education group | Weeks 6-7, Week 12, Weeks 18-19, Weeks 24-25
  Students will be randomized into Nudge intervention or Hygiene Education intervention at the completion of data collection in week 6, and the change in probability, or prevalence ratio, will be assessed over time, with measures at weeks 4-5, weeks 6-7, week 12, weeks 18-19 and weeks 24-25, comparing the probability of handwashing of nudge students post-toileting event to that of hygiene education students post-toileting event, measured using camera observations of the handwashing station outside of the latrine area.

SECONDARY OUTCOMES:
Change in the probability of handwashing with soap after a toileting event among students who received the early handwashing station intervention compared to students who received the late handwashing station intervention | Weeks 2-3, Weeks 4-5
  Students will be randomized into early handwashing station intervention (built in weeks 1-2) or late handwashing station intervention (built in weeks 3 and 4), and the change in probability, or prevalence ratio, will be assessed at week 2-3 and week 4-5, comparing the probability of handwashing of the early handwashing station students post-toileting event to that of the late handwashing station students post-toileting event, measured using camera observations of the handwashing station outside of the latrine area.
Change in the probability of handwashing with soap after a toileting event within the nudge intervention group, comparing students in the early handwashing station intervention to students in the late handwashing station intervention | Weeks 4-5, Weeks 6-7, Week 12, Weeks 18-19, Weeks 24-25
  In order to assess if the timing of the handwashing station building influences handwashing, the change in probability, or prevalence ratio, will be assessed over time, with observations at weeks 4-5, weeks 6-7, week 12, weeks 18-19 and weeks 24-25 within the Nudge group, comparing the probability of handwashing among students who received the early handwashing station (built in weeks 1 and 2) to the probability of handwashing among those students who received the late handwashing stations (built in weeks 3 and 4), measured using camera observations of the handwashing station outside of the latrine area.
Change in the probability of handwashing with soap after a toileting event within the hygiene education intervention group, comparing students in the early handwashing station intervention to students in the late handwashing station intervention | Weeks 4-5, Weeks 6-7, Week 12, Weeks 18-19, Weeks 24-25
  In order to assess if the timing of the handwashing station building influences handwashing, the change in probability, or prevalence ratio, will be assessed over time, with observations at weeks 4-5, weeks 6-7, week 12, weeks 18-19 and weeks 24-25 within the Hygiene Education group, comparing the probability of handwashing among students who received the early handwashing station (built in weeks 1 and 2) to the probability of handwashing among those students who received the late handwashing stations (built in weeks 3 and 4), measured using camera observations of the handwashing station outside of the latrine area.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hossain, Study Director — Save the Children; Mohini Venkatesh, Study Director — Save the Children; Pavani K Ram, MD, Study Director — University at Buffalo; Elise N Grover, MSPH, Study Director — University of Oklahoma; Robert Dreibelbis, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Save the Children, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Data on individual participants will not be shared.